CLINICAL TRIAL: NCT03513848
Title: Morning Light Treatment at Home to Reduce PTSD Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Alyson Zalta, Assistant Professor, Rush University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15122102
Record Dates: First submitted 2018-02-06; First posted 2018-05-02 (Actual); Results first posted 2019-10-23 (Actual); Last update posted 2019-10-23 (Actual); Status verified 2019-10

CONDITIONS: PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Bright Light (Experimental)
  Interventions: Device: Retimer
- Dim Light (Placebo Comparator)
  Interventions: Device: Retimer placebo

INTERVENTIONS:
Device: Retimer — The Retimer light device in this study is a commercially-available wearable light device. It permits ambulation while receiving light from LEDs positioned below the eyes. The LEDs emit green light (~500nm, 230 µW/m2, 500 lux), close to the peak sensitivity of circadian photoreceptors.
  Arms: Bright Light
Device: Retimer placebo — The Retimer device has been dimmed to reduce the light intensity to a level that will not shift circadian timing.
  Arms: Dim Light

SUMMARY:
There is evidence that some of the circadian photoreceptors, the intrinsically photosensitive retinal ganglion cells (ipRGCs), project directly to the amygdala, an area of the brain implicated in PTSD. Thus, a self-administered morning light treatment at home (shifts clock earlier and stimulates ipRGCs) may be a potentially efficacious adjunctive strategy for reducing PTSD symptoms. This study will test a 4 week daily 1 hour morning light treatment (active vs placebo) in individuals with PTSD. Outcome measures include measures of PTSD and depression.

ELIGIBILITY:
Inclusion Criteria:

* Probable PTSD based on the PCL-5 score
* Fluent in English
* Willingness and ability to comply with the protocol

Exclusion Criteria:

* Current or recent (past 6 months) alcohol or substance abuse problems
* Past or present psychotic or bipolar disorders
* Significant suicidal ideation or suicidal behaviors in past 6 months
* Unable or unwilling to give written informed consent.
* Severe hearing and memory problems.
* Cognitive impairment or mental retardation that interferes with subject being able to understand study requirements, consent form, etc.
* Special events (e.g. weddings, exams, surgery) planned during 5 weeks of study
* Unable to travel for study visits
* Pending legal cases/litigation
* Has a serious or unstable medical illness (including but not limited to cardiovascular disease, uncontrolled diabetes, advanced liver disease, kidney failure, seizures, cancer which is likely to result in hospitalization in next year).
* Reports significant chronic migraine. For migraines, subjects will only be excluded if they report that bright light can trigger migraines.
* Vision problems, retinal disease, or history of eye surgery.
* Taking photosensitizing medications
* Have previously had light treatment.
* Uncontrolled narcolepsy, sleep apnea or restless leg syndrome
* Likely to have undiagnosed, significant sleep apnea
* Likely to have undiagnosed, significant restless leg syndrome
* Prescribed hypnotics, over the counter sleep aids and antidepressants permitted providing all medications stable for 30 days before and during the study). All current medications must be non-photosensitizing.
* If in psychotherapy must have been for at least 30 days.
* People taking melatonin will be asked to abstain for a month before and during the study
* Has traveled outside the central time zone
* Have worked a night-shift the past month.
* Has winter depression
* Is pregnant, trying to get pregnant or breastfeeding.
* Household has a child <2 years old or a child that does not sleep through the night
* Is unavailable for a 5 week period
* Fail urine drug test at screening visit (after prescribed medication accounted for)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2018-06-27 (Actual); Study Completion 2018-06-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alyson Zalta, PhD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bright Light | Dim Light
Started | 9 | 6
Completed | 9 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bright Light | Dim Light | Total
Number analyzed (Participants) | 9 | 6 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.89 (9.36) | 51.00 (13.33) | 44.93 (11.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 5 | 2 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 4
  Not Hispanic or Latino | 6 | 5 | 11
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 5 | 8
  White | 4 | 0 | 4
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 9 | 6 | 15

OUTCOME MEASURES:

1. Primary Outcome: Change in PTSD Checklist for DSM-5 (PCL-5) Scores Over 4 Weeks of Treatment
Description: The PTSD Checklist for DSM-5 (PCL-5) is the gold standard measure of PTSD symptom severity. Range: 0-80. Higher scores indicate worse outcomes. We will assess change in PCL-5 scores over 4 weeks of treatment [Week 2 through Week 6 of the study].
Time Frame: Week 2 and Week 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bright Light | Dim Light
Number analyzed (Participants) | 9 | 6
units on a scale | 15.11 (14.38) | 2.50 (7.50)

2. Secondary Outcome: Change in Patient Health Questionnaire - 9 (PHQ-9) Scores Over 4 Weeks of Treatment
Description: The Patient Health Questionnaire - 9 (PHQ-9) is the gold standard measure of depression symptom severity. Range: 0-27. Higher scores indicate worse outcomes. We will assess change in PHQ-9 scores over 4 weeks of treatment [Week 2 through Week 6 of the study].
Time Frame: Week 2 and Week 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bright Light | Dim Light
Number analyzed (Participants) | 9 | 6
units on a scale | 4.78 (3.73) | 1.17 (5.95)

3. Other Pre Specified Outcome: Change in Sleep Duration Over 4 Weeks of Treatment
Description: Sleep duration will be captured using actigraphy data collected by the wrist actigraphy monitor worn by subjects throughout the intervention. We will assess change in sleep duration over 4 weeks of treatment [Week 2 through Week 6 of the study].
Time Frame: Week 2 and Week 6
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Change in Sleep Quality Over 4 Weeks of Treatment
Description: Sleep quality will be assessed using the Pittsburgh Sleep Quality Index (PSQI) with PTSD addendum. We will assess change in sleep quality over 4 weeks of treatment [Week 2 through Week 6 of the study].
Time Frame: Week 2 and Week 6
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over the 4 weeks of light treatment.
Arm/Group | Bright Light | Dim Light
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/6
Other Adverse Events (participants affected / at risk) | 1/9 | 0/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bright Light (N=9) | Dim Light (N=6)
Headache (Nervous system disorders) | 1 (1) | 0 (0) — Mild headache

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-19): https://cdn.clinicaltrials.gov/large-docs/48/NCT03513848/Prot_SAP_001.pdf